CLINICAL TRIAL: NCT01261377
Title: Comparison of Effects of Bi-level Positive Airway Pressure Therapy and Nocturnal Oxygen Therapy on Right and Left Ventricular Hemodynamics in Overlap Syndrome (Co-existent Chronic Obstructive Airway Disease and Obstructive Sleep Apnea)
Brief Title: Cardiac Hemodynamics in Overlap Syndrome (COPD With Obstructive Sleep Apnea)
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: the fellow interested in this project left the institution
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Atul Malhotra, MD, Atul Malhotra, MD, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-P001753
Record Dates: First submitted 2010-12-15; First posted 2010-12-16 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Chronic Obstructive Airway Disease
Keywords: COPD, obstructive sleep apnea, OSA, BPAP, CPAP
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Sleep Apnea, Obstructive; Microcephaly, Primary Autosomal Recessive, 6 | interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Bi-level positive airway pressure (BPAP) (Active Comparator): bi-level will be titrated to optimize oxygenation and ventilation.
  Interventions: Device: Bi-level positive airway pressure (BPAP)
- Nocturnal oxygen (Active Comparator): oxygen will be provided as per standard of care.
  Interventions: Drug: Oxygen
- Continuous positive airway pressure (Active Comparator): The level of CPAP will be titrated to treat OSA. The duration of therapy will be six months.
  Interventions: Device: CPAP

INTERVENTIONS:
Device: Bi-level positive airway pressure (BPAP) — The level of BPAP will be titrated to treat OSA as well as hypoxemia and hypercapnia. The duration of therapy will be six months.
  Arms: Bi-level positive airway pressure (BPAP)
Drug: Oxygen — Oxygen will be titrated to keep resting oxygen saturation (as measured by pulse oximeter) more than 88 percent. The duration of therapy will be six months.
  Arms: Nocturnal oxygen
Device: CPAP — The level of CPAP will be titrated to treat OSA. The duration of therapy will be six months.
  Arms: Continuous positive airway pressure

SUMMARY:
Patients with both sleep apnea and COPD have overlap syndrome, but their optimal management is not known. We plan to conduct a randomized trial of of bi-level PAP vs. night time oxygen to asses the impact of intervention on cardiac MRI and biomarkers.

DETAILED DESCRIPTION:
Presence of chronic obstructive pulmonary disease (COPD) and obstructive sleep apnea (OSA) in the same patient has been termed overlap syndrome, affecting 1% of the U.S. population. Despite the high prevalence of overlap syndrome, little research has been done in this field. Overlap syndrome has been recently reported to have higher death rate than COPD alone, which is due to effect on the heart. However, the mechanisms by which overlap syndrome affects the heart are not known well. Also, the ideal treatment for overlap syndrome is not known.

This study is being done to find the mechanisms by which overlap syndrome affects the right and left sides of heart (using cardiac MRI to study the heart). We will also compare the effect of treatment with bi-level positive airway pressure device (BPAP) vs. night-time oxygen on heart in overlap syndrome. These aims will allow us to test the hypothesis that overlap syndrome patients have worse heart function than COPD only or OSA only, and treatment with BPAP device will improve the heart function better than oxygen only.

At the baseline visit, the subject will undergo an overnight sleep study in the hospital. In the morning, blood draw to measure serum inflammatory biomarkers (C-Reactive Protein, interleukin-6, P-selectin, ICAM-1, TNF-alpha), urine catecholamine level, six-minute walk test, questionnaire for health-related quality of life score and modified Medical Research Council (MMRC) dyspnea score, lung function tests, ultrasound of forearm blood vessels and cardiac MRI will be done. No follow-up visit is needed if the subject does not have sleep apnea. If the subject has sleep apnea based on the sleep study, he/she will be allotted to treatment with a BPAP device or night-time oxygen for 6 months. If the subject does not want to be treated with BPAP or oxygen, CPAP device will be used to treat sleep apnea. During the duration of study treatment, phone calls and a brief study visit at 3 months will be done to make sure there is no discomfort related to the treatment. After 6 months of study treatment, cardiac MRI, ultrasound of forearm blood vessels, lung function tests, blood draw for serum inflammatory biomarkers, urine catecholamine level, six-minute walk test, and questionnaires for dyspnea score and quality of life score will be repeated.

This study will help us in better understanding of mechanisms of high death rate due to effects on the heart in overlap syndrome. It will also help us in understanding better ways to treat sleep apnea in COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Both men and women with age more than 18 years.
* Known diagnosis of COPD (GOLD stage 2 or higher).

Exclusion Criteria:

* Already using CPAP or BPAP device.
* Estimated GFR <30 ml/min/1.73 m2 or on hemodialysis.
* Women known to be pregnant or planning to be pregnant in next 6 months.
* Cardiac pacemaker, metallic heart valves, metallic implants, claustrophobic.
* Chronic atrial fibrillation or frequent premature ventricular contractions.
* Using lipid-lowering medications, aspirin, oral steroids, steroid-sparing medications or anti-oxidant vitamin supplements.
* If taking sildenafil or related drugs, unable to stop it within 48 hours of the study visit.
* Contraindications to stress cardiac testing: acute myocardial infarction within 48 hours, unstable angina not yet stabilized with medical therapy, ongoing chest pain, active broncho-constriction, uncontrolled cardiac arrhythmia, symptomatic severe aortic stenosis, aortic dissection, acute pulmonary embolism or pericarditis.
* Uncontrolled COPD or acute COPD exacerbation.
* Known chronic inflammatory diseases like lupus or active infection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-11; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Right ventricular end-diastolic volume | Six months

SECONDARY OUTCOMES:
Other cardiac hemodynamics parameters (end-systolic volume, ejection fraction, mass index and wall motion of right and left ventricles, coronary blood flow, pulmonary artery pressure and blood flow, etc.) | Six months
Serum inflammatory biomarkers (C-reactive protein, interleukin-6, ICAM-1 and P-selectin) | Six months
Urine catecholamine level | Six months
Flow mediated dilatation of brachial artery | Six months
Pulmonary Function tests | Six months
BODE Index | Six months

CONTACTS AND LOCATIONS:
Overall Officials: Atul Malhotra, MD, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Massachussets General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No
nothing to include